CLINICAL TRIAL: NCT05399108
Title: Ultrasound-guided Vena Jugularis Interna Catheterization Lateral Approach Short Axis in - Plane Technique
Brief Title: Ultrasound Guided Vena Jugularis Interna Catheterization Lateral Approach Short Axis in - Plane Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masarykova Nemocnice v Usti nad Labem, Krajska Zdravotni a.s. (Other)
Responsible Party: Principal Investigator, Michal Kalina, Principal Investigator, Masarykova Nemocnice v Usti nad Labem, Krajska Zdravotni a.s.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UltrasoundLateralCannulation
Record Dates: First submitted 2022-05-23; First posted 2022-06-01 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Central Vein Catheter
Keywords: ultrasound guided catheterization; central vein catheterization; jugular vein catheterization; in-plane catheterization

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Novel Lateral Approach (Experimental): In this arm, the catheterization of the internal jugular vein is done with ultrasound guidance displaying the vein on its short axis using a lateral approach and in-plane technique. The catheterization is done according to the newest international recommendations for good clinical practice.
  Interventions: Procedure: Ultrasound Guided Lateral Approach Catheterization of Jugular Internal Vein
- The Conventional Approach (Active Comparator): In this group catheterization of the jugular internal vein is done by conventional approach with ultrasound guidance using displaying on its short axis and using the out-of-plane technique.
  Interventions: Procedure: Ultrasound Guided Conventional Approach Catheterization of Jugular Internal Vein

INTERVENTIONS:
Procedure: Ultrasound Guided Lateral Approach Catheterization of Jugular Internal Vein — The jugular internal vein is displayed on its short axis. On the image are displayed the trapezius muscle and layers of skin. Just above the trapezius muscle using the in-plane technique is done puncture of the vein. By Seldinger's technique, catheterization is done. The whole procedure is done according to the newest international recommendations for central vein catheterization.
  Arms: The Novel Lateral Approach
Procedure: Ultrasound Guided Conventional Approach Catheterization of Jugular Internal Vein — The jugular internal vein is displayed on its short axis. The cannulation is done by the conventional approach (middle approach - the most frequently used).
  Arms: The Conventional Approach

SUMMARY:
Central venous access is one of the most frequently used venous accesses in intensive care units. Insertion of the central venous catheter belongs to the basic skills of an intensivist. One of the veins that are available for catheterization is the internal jugular vein. It is recommended to perform jugular vein catheterization along with real-time ultrasound guidance.

Imaging of the jugular vein is usually performed in two ways: on the short axis or on the long axis. The puncture method is described based on the type of needle imaging technique, out-of-plane or in-plane method.

Traditionally, catheterization is performed by a medium approach during imaging the vein on a short axis using the out-of-plane technique. The main advantage of this procedure is proper imaging of the jugular vein and surrounding anatomical structures. However, the limited needle display is rather inconvenient, as only the needle tip can be displayed. This method of central venous catheterization has a first attempt success rate of 80%.

This study is going to concentrate on discussing the performing of jugular vein catheterization by a novel lateral approach in-plane technique during imaging of the vein on the short axis. This procedure for placement of a central venous catheter into the internal jugular vein has not yet been described nor investigated. The above-mentioned method combines the advantage of reliable jugular vein imaging together with proper imaging of the whole needle. At the same time, the fixation of the catheter in the supraclavicular region allows for a better nursing routine, hence increasing the patient's comfort.

DETAILED DESCRIPTION:
All potential candidates to enroll will undergo an examination by an anesthetist. If the candidate meets inclusion/ exclusion criteria, the candidate will sign an informed consent and be enrolled in the study. The calculated number of needed subjects is 180 (90 in each group). In the next step, all enrolled subjects will be randomized by computer block randomization into two groups.

* In group A catheterization of vena jugularis interna will be done by lateral approach with visualization of the vein on its short axis with ultrasound and the in-plane technique will be used.
* In group B catheterization of the vena jugularis interna will be done by conventional approach with visualization of the vein on its short axis with ultrasound and the out-of-plane technique will be used.

Later then all enrolled subjects will undergo examination by an anesthetist or neurologist focused on neurological deficits in the upper limbs. The assessment will be done by Neurological Impairment Scale (NIS).

In the next step catheterization of the vein will be done according to the latest international recommendations and the randomized group.

The time of the start of catheterization and the time of the end of catheterization will be recorded.

On daily basis, there will be done function control of the central vein catheter. The control is done by aspiration from all accesses. Unproblematic aspiration from all accesses will be interpreted as a functional catheter.

On daily basis, there will be done ultrasound control of the catheter to evaluate the presence of thrombosis.

On daily basis, there will be control of the insertion site of the catheter any complications such as signs of an infection or signs of catheter damage will be recorded.

Before extraction of the catheter, there will be examined by an anesthetist or neurologist to evaluate neurological impairment in the upper limbs. The reason and the date of the extraction of the catheter will be recorded.

All measured data will be recorded on the case report form and also will be recorded in the patient's hospital medical documentation. The recorded data will be processed by standard statistical tests such as T-tests and students test.

The aim of this study is to prove the noninferiority of the novel lateral approach.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years with an indication of central venous catheter placement

Exclusion Criteria:

* Not signing the informed consent
* BMI under 16,5
* Contraindication of central venous catheter placement into internal jugular vein (thrombosis, site infection, bleeding diseases, anticoagulation or antiaggregation therapy)
* hypersensitivity to sterile ultrasound gel
* neurological impairment on upper limbs
* neurodegenerative disorder

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Success rate of first attempt | Measured from the time the cannulation starts (local anesthetic infiltration) till insertion of the catheter, up to 120 minutes.
  Primary outcome is to prove that first attempt success rate by the novel approach is comparable with the success rate of the first attempt success rate of the conventional approach.

SECONDARY OUTCOMES:
Rate of complications | Measured from the start of cannulation (local anesthetic infiltration) till extraction of the catheter, up to 45 days.
  Secondary outcome is to prove that rate of complications between both approaches the novel one and the conventional one are comparable.
Risk of neurological impairment assessed by Neurological Impairment Scale | Measured from insertion the catheter till the extraction of the catheter, up to 45 days.
  Secondary outcome is to prove that risk of developing new neurological impairment is comparable between the novel approach and the conventional approach. We will assess the neurological impairment by Neurological Impairment Scale. This scale identify whether there is or there is not neurological impairment and distinguish between motor or sensory impairment. Maximum points for one upper limb if five. Minimum points for upper lim is zero. Zero points means there is no neurological impairment. Five points means there is neurological impairment in all segments from C5 to T1.
Functional time of the catheter | Measured from inserting the catheter till the extraction of the catheter, up to 45 days.
  Secondary outcome is to prove that functional time of the catheter is comparable between the novel approach and the conventional approach.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Kalina, MUDr., Principal Investigator — Krajská Zdravotní a.s. Masarykova Nemocnice v Ústí nad Labem
Locations (1):
- Masarykova Nemocnice v Ústí nad Labem, Krajská Zdravotní a.s., Ústí nad Labem, Ústí Nad Labem Region, Czechia

IPD SHARING:
Plan to Share IPD: No